CLINICAL TRIAL: NCT00865033
Title: A Relative Bioavailability Study of Metformin HCL 1000 mg Tablets Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of Metformin HCL Tablets, 1000 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B053709
Record Dates: First submitted 2009-03-15; First posted 2009-03-19 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

ARMS (2):
- 1 (Experimental): Metformin HCL Tablets, 1000 mg
  Interventions: Drug: Metformin HCL Tablets, 1000 mg Sandoz
- 2 (Active Comparator): Glucophage 1000 mg Tablets
  Interventions: Drug: Glucophage 1000 mg

INTERVENTIONS:
Drug: Metformin HCL Tablets, 1000 mg Sandoz
  Arms: 1
Drug: Glucophage 1000 mg
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioequivalence of Metformin HCL Tablets, 1000 mg under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services